CLINICAL TRIAL: NCT01139710
Title: Sarcoidosis-associated Pulmonary Hypertension
Status: Completed | Type: Observational
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC10-114-10.CTIL
Record Dates: First submitted 2010-06-07; First posted 2010-06-08 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2011-07

CONDITIONS: SARCOIDOSIS
Keywords: SARCOIDOSIS; PULMONARY HYPERTENSION; outpatients clinic at Meir medical center
MeSH Terms: conditions — Sarcoidosis; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective study was conducted to explore clinical characteristics and outcomes of patients diagnosed with pulmonary sarcoidosis and PH. The investigators also assessed the role of D -dimer levels in these population.

DETAILED DESCRIPTION:
The investigation will be approving by the Ethics Committee of Meir medical center.

We retrospectively will review the medical records of 100 sarcoidosis patients seen in our outpatient pulmonary clinics of Meir medical center, between July 2009 and May 2010.

All the patients will prospectively invite to our pulmonary outpatients clinic at Meir medical center.

Sarcoidosis will be diagnosed based on the latest American Thoracic Society (ATS), European Respiratory Society (ERS) and World Association of Sarcoidosis and Other Granulomatous Disorders (WASOG) criteria. (6, 7) Each patient will undergo two-dimensional echocardiographic data, complete pulmonary function test results including spirometry, lung volume, CO diffusion capacity and 6-min walk test (6MWT) data and D-dimer assay during their visiting.

Data will be collecting including patient demographics, symptoms, details of comorbid illnesses, sarcoidosis stage using the modified Scadding (8) classification system to stage chest radiography (CXR) findings and treatment.

Pulmonary function tests included spirometry and lung volume measurement by body plethysmography, performed according to the recommendations of the American Thoracic Society. (9) The 6MWT was conducted in accordance with ATS guidelines. (10) All patients exhibited resting oxygen saturation (SpO 2 ) the > 88% at the beginning of the walk test and Borg dyspnea index (11) will be record at the beginning and end of the 6-min walk.

All Computed tomography (CT) findings of the patients will be assess for the presence of the following recognized CT patterns (12): (1) mediastinal and/or hilar lymph node enlargement; (2) ground-glass opacity; (3) consolidation; (4) nodules <3 cm in diameter; (5) thickening of bronchovascular bundles; (6) linear opacity, including interlobular septal lines and interstitial thickening and (7) features indicating scarring and fibrosis (grouped together) that included traction bronchiectasis, honeycombing, cysts and/or volume loss.

In addition, all CT will be review for findings that are known as a signs of PH including the pulmonary trunk diameter, right and left pulmonary arteries diameters and the pulmonary to aortic diameters ratio.

The radiologist will be blinded to the echocardiological data as well as to the pulmonary function data and D-dimer levels.

Diagnosis of PH was based on Doppler echocardiography and defined as an estimated right ventricular systolic pressure (RVSP) of the > 40 mm Hg in the absence of left ventricular dysfunction (i.e., an ejection fraction under 50%), ischemic heart disease (manifested by regional wall motion abnormalities) or valvular heart disease. Right ventricular systolic pressure was estimated based on the modified Bernoulli equation (13) RVSP = transtricuspid gradient + right atrial pressure (RAP), where transtricuspid gradient is 4v2 (v = peak velocity of tricuspid regurgitation in meter per second) and RAP was estimated to be 5, 10 All the patients will undergo a D-dimer assay in the same day of the pulmonary function tests and Echo evaluations.

ELIGIBILITY:
Inclusion Criteria:

* All patients above 18 years old

Exclusion Criteria:

* Non sarcoidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 sarcoidosis patients
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
to explore clinical characteristics and outcomes of patients diagnosed with pulmonary sarcoidosis and PH | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Meir MC, Kfar Saba, Israel, Israel